CLINICAL TRIAL: NCT00757562
Title: Multiple-Dose Safety and Tolerance Study of Desloratadine in Atopic Pediatric Subjects and Pediatric Subjects With Chronic Idiopathic Urticaria, Ages >=2 to <12 Years, Who Are Poor Metabolizers of Desloratadine
Brief Title: Safety of Desloratadine in Children With Allergy Sensitivity and Chronic Hives, Who Are Poor Metabolizers of Desloratadine (Study P02994)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P02994
Expanded Access: Available
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Chronic Idiopathic Urticaria; Atopy
MeSH Terms: conditions — Chronic Urticaria | interventions — desloratadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DL (Experimental): Desloratadine syrup once daily
  Interventions: Drug: desloratadine
- Placebo (Placebo Comparator): placebo syrup once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: desloratadine — desloratadine syrup: 1.25 mg (2.5 mL) for subjects >=2 to <6 years, 2.5 mg (5 mL) for subjects >=6 to <12 years, orally once daily in the morning for 36 days.
  Other Names: SCH 034117; Clarinex
  Arms: DL
Drug: Placebo — placebo syrup: 2.5 mL for subjects >=2 to <6 years, 5 mL for subjects >=6 to <12 years, orally once daily in the morning for 36 days.
  Arms: Placebo

SUMMARY:
This study was conducted to evaluate the safety and tolerance of desloratadine after 5 weeks of repetitive dosing in children ages 2 to 12 years old with allergic hypersensitivity or chronic hives. All of the subjects enrolled in this trial were previously identified in an earlier trial to be poor metabolizers of desloratadine.

ELIGIBILITY:
Inclusion Criteria:

Subjects must:

* have been previously identified through the previous study P03031 to be atopic or with chronic idiopathic urticaria and be a poor metabolizer of desloratadine.
* have clinical laboratory tests within normal limits.
* be in good health, free of any clinically significant disease that could interfere with the study.
* normal 12-lead ECG

Exclusion Criteria:

Subjects who:

* have a history of any clinically significant local or systemic infectious disease within 4 weeks prior to treatment.
* have taken any medication that is restricted by the protocol or failed to satisfy washout requirements.
* are allergic to desloratadine.
* have used a loratadine- or desloratadine-containing product within the past 30 days.
* are female and menstruating.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2002-11-01 (Actual); Primary Completion 2003-10-01 (Actual); Study Completion 2003-10-01 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerance | Weekly throughout the 5-week study (Day 1, Day 8, Day 15, Day 22, Day 29, and Day 36).

SECONDARY OUTCOMES:
Plasma concentration data (of desloratadine to loratadine) prior to administration of desloratadine on Days 15 and Days 36. | Days 15 and Days 36